CLINICAL TRIAL: NCT04850469
Title: Study of Exosomes Derived From Mesenchymal Stem Cells on the Therapy for Children With Severe Infection
Brief Title: Study of MSC-Exo on the Therapy for Intensively Ill Children
Status: Withdrawn | Type: Observational
Why Stopped: Lacking of funding
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-13
Record Dates: First submitted 2021-03-26; First posted 2021-04-20 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Sepsis; Critical Illness
Keywords: Sepsis; Critical Illness; Mesenchymal Stem Cell Derived Exosomes
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- trial group: Mesenchymal Stem Cell-Derived Exosomes
- control group: conventional treatment

SUMMARY:
At present, a number of projects related to MSCs have been approved for graft-versus-host disease, myocardial infarction, Crohn's disease and other diseases, indicating a strong therapeutic potential of MSCs. However, the efficacy of MSC-Exo for severely infected children is not fully evaluated. In our study, patients who met the inclusion criteria will be divided into trial group and control group. Clinical and demographic data, as well as treatment outcome will be collected from the electronic health record. This study will evaluate the application and therapeutic effect of MSC-Exo in severely infected children, and determine the Optimal dosage and infusion.

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSCs) are pluripotent stem cells with high self-renewal ability and multidirectional differentiation potential. studies revealed that local or systemic administration of mesenchymal stem cell-derivrd exosomes (MSC-Exo) efficiently suppressed detrimental immune response in inflamed tissues and promoted survival and regeneration of injured parenchymal cells. European Union countries have written MSCs into treatment guidelines for refractory graft-versus-host disease.

In China, the technology for isolation, in vitro culture and expansion of MSCs is already mature. With further research on the therapeutic efficacy of MSC-Exo and the development of clinical trials, it is expected to become a treatment for severe illness.

A predictable infection plan is going to be widely used in clinics to provide individualized treatment for patients, improve the prognosis of patients and improve the quality of life.

The investigators intend to enroll all children who were hospitalized in pediatric intensive care unit PICU of Children's Hospital of Fudan University from January 2022 to December 2023. Children with a PICU length of day less than 48h will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* children hospitalized in PICU of Children's Hospital of Fudan University

Exclusion Criteria:

* discharge within 48 hours
* patients without informed consent
* incomplete clinical and demographic data

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children hospitalized in PICU of Children's Hospital of Fudan University from January 2022 to December 2023
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The death rate of children | within 28 days after they discharged from PICU
  The death rate of children in 28 days after their discharged from PICU
Marshall Multiple Organ Dysfunction Score | Within 3 to 15 days after the start of treatment
  The Marshall Multiple Organ Dysfunction Score (MODS) assesses the same six organ systems using slightly different values for four grades of organ dysfunction. The total score, ranging from 0 to 24, arises from the sum of all single organ scores using the first measured value of the day. Intervals for the most abnormal value of each variable were constructed on a scale from 0 to 4 so that a value of 0 represented essentially normal function and was associated with an ICU mortality rate of < 5%, whereas a value of 4 represented marked functional derangement and an ICU mortality rate of > or = 50%.
the APPS score | Within 3 to 15 days after the start of treatment
  The APPS is a 9-point score that is calculated by measuring the age, PaO2/FIO2 ratio, and plateau pressure at 24 h after the patient is diagnosed with moderate to severe ARDS and counting each one to 1-3. Since many variables are not needed for calculations, clinicians can easily predict the in-hospital mortality of mechanically ventilated patients with moderate to severe ARDS patients at bedside.

SECONDARY OUTCOMES:
length of stay in PICU | up to 28 days
  Time from PICU admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Lu, Doctor, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China